CLINICAL TRIAL: NCT00123942
Title: Phase I Trial of MEDI-507 in CD2-Positive Lymphoproliferative Disease
Brief Title: Trial of MEDI-507 in CD2-Positive Lymphoproliferative Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After review of safety events and have decided that further dose escalation of MEDI-507 as a single agent is not feasible.
Sponsor: MedImmune LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP099; NCT00071825 (obsolete NCT alias); NCT00075361 (obsolete NCT alias)
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Lymphoproliferative Disorders
Keywords: CD2+ Lymphoproliferative disorder
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — siplizumab

INTERVENTIONS:
Drug: MEDI-507

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) and safety and tolerability of MEDI-507 in patients with CD2-positive lymphoproliferative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age. Women of childbearing potential must have a negative serum pregnancy test within 5 days of the initial MEDI-507 administration and a negative urine pregnancy test on Day 0 prior to receiving the first dose of MEDI-507. Women of childbearing potential must agree to practice an effective method of contraception. Sexually active males must agree to use a condom.
* Histologically confirmed diagnosis of a lymphoproliferative disorder as determined by the Laboratory of Pathology at the Clinical Center at the National Institutes of Health (NIH). Only patients with the following lymphoproliferative disorders will be eligible:

  * ATL: Patients with all except the smoldering form of adult T-cell leukemia/lymphoma (ATL) will be eligible, regardless of whether they have had previous therapy, since there is no effective standard of care therapy for this disease;
  * CTCL: Patients with all stages of cutaneous T-cell lymphoma (CTCL) are eligible with the exception of Stage Ia. Patients with Stages Ib through III are eligible if their disease has failed at least one standard form of prior therapy;
  * PTCL: Patients with Stages I-IV peripheral T-cell lymphoma (PTCL) are eligible if their disease has progressed after standard chemotherapy;
  * LGL: Patients with large granular lymphocyte leukemia (LGL) must have myelosuppression (granulocyte count ≤1,500/uL; platelet count ≤75,000/uL; or hemoglobin ≤10 g/dL), or require hematopoietic support (transfusion or colony stimulating factors including filgrastim, IL-11, or erythropoietin) to maintain counts at these or higher levels or systemic symptoms (fever, night sweats or weight loss). Patients must have disease that is unresponsive to one prior therapy. Patients with monoclonal and polyclonal forms of the disease will be eligible.
* Cells must express CD2. CD2 expression will be verified by immunohistochemistry in the Laboratory of Pathology at the NIH. At least 30% of tumor cells must be CD2 positive for the patient to be eligible for the study by immunohistochemistry. CD2 staining will be performed on existing tissue blocks and on fresh tumor tissue if a biopsy is performed. It is expected that the majority of patients will have CD2 expression evaluated by flow cytometry and the majority of cells will express the marker.
* Measurable or evaluable disease.
* Karnofsky Performance Status ≥70%.
* Life expectancy of >2 months.
* Granulocyte count ≥1,000/mm3 and a platelet count ≥50,000/mm3. Patients with LGL leukemia are excluded from these criteria. For patients with LGL leukemia, ANC and platelet count will not be considered in determining study eligibility.
* Serum creatinine <1.5 mg/dL.
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) value ≤2.0-fold greater than the upper limit of normal (if due to lymphoma in the liver, patients will be allowed to have transaminase values ≤ 5.0 fold greater than the upper limit of normal) and bilirubin ≤2.0 mg/dL unless due to Gilbert's syndrome (unconjugated hyperbilirubinemia) in which case the bilirubin should be ≤3.5 mg/dL.
* Prior treatment with cytotoxic chemotherapy, surgery, and prolonged cytolytic steroid therapy is allowed provided last treatment was given at least 3 weeks prior to first dose of study drug administration and all toxicities have resolved.
* Prior treatment with other investigational anticancer drugs and monoclonal antibodies is allowed provided the last treatment was given at least 30 days prior to the first dose of study drug administration.
* Patients must understand and sign a National Cancer Institute (NCI) pre-screening consent form and a protocol specific informed consent form prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

* Known history of central nervous system (CNS) disease.
* Pregnant or nursing. The effects of MEDI-507 on the developing fetus and the nursing infant are unknown.
* Positive for human immunodeficiency virus (HIV) because of the risk of increased HIV-associated complications due to increased immunosuppression.
* Positive for hepatitis B surface antigen or with antibodies to hepatitis C virus because the therapy may be associated with increased viral replication.
* Symptomatic CMV positivity or CMV PCR >1000 copies
* Prior treatment with MEDI-507.
* Prior history of significant adverse events related to previously administered monoclonal antibody.
* History within 6 months prior to first dose of study drug administration or evidence of intercurrent illnesses including myocardial infarction, uncontrolled hypertension, stroke, or transient ischemic attacks.
* Respiratory insufficiency requiring oxygen therapy or O2 saturation less than 90% by pulse oximetry.
* Active infection requiring systemic anti-infective therapy or other physical or psychological illnesses that would increase risk to the patient, in the opinion of the Principal Investigator.
* Any general medical or psychological or behavioral conditions that, in the opinion of the investigator, may pose additional risk in administering study drug to the patient or will not permit the patient to complete the study or sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2004-04

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) or the optimal biological dose
(OBD) of MEDI-507 based on safety and tolerability of MEDI-507 in patients with
CD-2 positive lymphoproliferative disorders.

CONTACTS AND LOCATIONS:
Overall Officials: John Janik, MD, Principal Investigator — National Cancer Institute (NCI); Karen Kaucic, MD, Study Director — MedImmune LLC
Locations (1):
- National Cancer Institute/National Institutes of Health, Bethesda, Maryland, United States